CLINICAL TRIAL: NCT06961019
Title: A Proof-of-Science, Single-Treatment, Two-Group, Clinical Evaluation of Safety, In-Use Tolerability, Efficacy of Herbal-Based Sugar Support Effervescent Tablets in Type-2 Diabetes Mellitus (T2DM) Patients
Brief Title: Clinical Study to Assess the Safety, Efficacy and In-Use Tolerability of Herbal-Based Sugar Support Effervescent Tablets in Type-2 Diabetes Mellitus Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NovoBliss Research Pvt Ltd (Other)
Collaborators: Zywie Ventures Private Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NB250012-ZV
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Type2 Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Arm Sugar support effervescent Tablets (Experimental): T2DM patients who are on treatment of 500mg Metformin dose. Test Product Name: Sugar support effervescent tablets Product By: Zywie Ventures Private Limited. Mode of Usage: Dissolve one effervescent tablet in a full glass of water (approximately 200 mL). Allow it to fully dissolve before consuming. For best results, consume the solution immediately after preparation. Frequency: Twice a day before the meal Route of Administration: Oral
  Interventions: Other: Sugar support effervescent Tablets
- Test Arm Placebo (Experimental): T2DM patients who are not on medication and Diabetes Mellitus managed by only dietary/herbal supplements and exercise . Test Product Name: Sugar support effervescent tablets Product By: Zywie Ventures Private Limited. Mode of Usage: Dissolve one effervescent tablet in a full glass of water (approximately 200 mL). Allow it to fully dissolve before consuming. For best results, consume the solution immediately after preparation. Frequency: Twice a day before the meal Route of Administration: Oral
  Interventions: Other: Sugar support effervescent Tablets

INTERVENTIONS:
Other: Sugar support effervescent Tablets — Dissolve one effervescent tablet in a full glass of water (approximately 200 mL). Allow it to fully dissolve before consuming. For best results, consume the solution immediately after preparation.
  Frequency: Twice a day before the meal Route of Administration: Oral

SUMMARY:
This is a Proof-of-Science, exploratory, prospective, single-treatment, two-group, clinical safety, efficacy and tolerability study of herbal based Sugar support effervescent tablets on the patients with Type 2 Diabetes Mellitus.

DETAILED DESCRIPTION:
A total of 14 male and non-pregnant |non-lactating female (7 patients managing diabetes with 500 mg Metformin dose and 7 patients managing by only dietary/ herbal supplements and exercise) with the age of 18-65 years will be enrolled to complete 12 subjects (6 patients managing diabetes with 500 mg Metformin dose and 6 patients managing by only dietary/ herbal supplements and exercise) the study. A sufficient number of patients will be pre-screened based on HbA1c (6.5% to 8% gm) levels to ensure that enough subjects successfully qualify the screening. The potential subjects will be screened on the basis of the inclusion and exclusion criteria only after obtaining the written informed consent from the subjects. Subjects will be pre-screened by the screening department of NovoBliss Research. Subjects will be called telephonically by the recruiting department prior to the enrolment visit. The subject will be asked to bring the past medications, or laboratory reports along with on the study visit day. The subjects will be instructed to visit the facility as per the below visits:

Visit 01 (Within 15 Days from Day 01): Screening, Baseline Evaluation Visit 02 (Day 01): Enrolment, Test Treatment Starts Visit 03 (Day 30 + 2 Days): Evaluation, Test Treatment phase Visit 04 (Day 60 + 2 Days): Evaluation, Test Treatment phase Visit 05 (Day 90 + 2 Days): Final Evaluations, End of the study

ELIGIBILITY:
Inclusion Criteria:

* 1) Male and female individuals with the age between 18 to 65 years at the time of consent.

  2) Subject diagnosed with T2DM. 3) Subjects with currently having HbA1c values between 6.5% to 8.0 gm%. 4) Subjects currently managing T2DM by dietary or herbal supplements and exercise only for at least 8 weeks prior to screening for Group 1.

  5) Subjects currently managing T2DM by 500 mg Metformin dose for Group 2. 6) Subjects having prescription or diabetes related laboratory reports at the time of screening.

  7) Subjects willing to come in fasting state for every study visit. 8) Subjects are willing to give written informed consent and are willing to come for regular follow up.

  9) Subjects who commit not to use other medications other than the allocated test treatment for the entire duration of the study.

  10) Subjects who have note participated in any other similar clinical study in last 3 months.

  11) Willing to use test treatment throughout the study period.

Exclusion Criteria:

* 1) Subjects diagnosed with other types of Diabetes like T1DM or specific type of DM (i.e., pancreatic injury induced DM, diabetes mellitus caused by Cushing's syndrome or acromegaly, Latent Autoimmune Diabetes in Adults (LADA), Maturing Onset diabetes of the young (MODY) etc.) 2) Subjects with any end organ damage due to diabetes (including microvascular complications like retinopathy, nephropathy and macrovascular complications like ischemic heart disease, peripheral vascular disease and cerebrovascular disease resulting in organ and tissue damage) within 6 months prior to screening.

  3) Subjects taking any weight loss medication or dietary supplements, have participated in a weight loss program within 4 weeks prior to screening.

  4) Subjects taking any glucose modifying medication like Sulfonylureas, Biguanides (Except 500 mg Metformin), Meglitinides, Thiazolidinediones, DPP-4 inhibitors, GLP-1 agonist, SGLT2 inhibitor, Alpha-glycosidase inhibitors or any other within 8 weeks prior to screening.

  5) Subjects having history of drug or alcohol use. 6) Subjects having history of smoking or currently smoking or using any form of smokeless tobacco.

  7) Subjects who have deviations in the laboratory reports which could warrant exclusion from the study, as per investigator's opinion.

  8) Individuals with uncontrolled hypertension defined as Systolic blood pressure ≥ 140 mm Hg and/or Diastolic blood pressure ≥ 90 mm Hg with or without anti-hypertensives.

  9) Subjects who are hypersensitive to any of the components of the treatment. 10) Subjects who have planned major changes in the lifestyle (i.e., diet, dieting, exercise level, significant travel) during the duration of the study.

  11) Participation in a study of any other treatment within 90 days prior to the screening.

  12) Pregnant or breastfeeding or planning to become pregnant during the study period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-03-14 (Estimated); Study Completion 2026-03-14 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1C values | Before administration on Day 01 and post dose on Day 90
  To evaluate the effectiveness of the test treatment in terms of change in HbA1C values
Change in FBG level | Before administration on Day 01 and post dose on Day 30, Day 60 and Day 90
  To evaluate the effectiveness of the test treatment in terms of change in FBG Level
Change in PPBG level | Before administration on Day 01 and post dose on Day 30, Day 60 and Day 90
  To evaluate the effectiveness of the test treatment in terms of change in PPBG level

SECONDARY OUTCOMES:
Change in body weight using by using calibrated weighing balance | Before administration on Day 01 and post dose on Day 30, Day 60 and Day 90
  To evaluate the effectiveness of the test treatment in terms of change in body weight
Change in waist to hip circumference by using calibrated measuring tape | Before administration on Day 01 and post dose on Day 30, Day 60 and Day 90
  To evaluate the effectiveness of the test treatment in terms of change in the waist to hip circumference
Change in BMI | Before administration on Day 01 and post dose on Day 30, Day 60 and Day 90
  To evaluate the effectiveness of the test treatment in terms of change in BMI
Change in Satiety score by VAS scoring scale | Before administration on Day 01 and post dose on Day 30, Day 60 and Day 90
  To evaluate the effectiveness of the test treatment in terms of change in satiety (10- High Satiety Level and 1- Low satiety level)
Chane in quality of life by Short Form Health Survey (SF-36) | Before administration on Day 01 and post dose on Day 30, Day 60 and Day 90
  To evaluate the effectiveness of the test treatment in terms of change in Quality-of-life questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Nayan Patel, MBBS, Principal Investigator — NovoBliss Research Private Limited
Locations (1):
- NovoBliss Research Pvt Ltd, Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No